CLINICAL TRIAL: NCT02077803
Title: A Single-Dose, Open-Label, Randomized, 3-Way Crossover Pivotal Study to Assess the Bioequivalence of the Fixed Dose Combination Tablets of Canagliflozin and Metformin Extended Release (XR) (2 x 50 mg/1,000 mg) With Respect to the Individual Components of Canagliflozin (1 x 100 mg) and Metformin XR Tablet (4 x 500 mg) in Healthy Fed Subjects
Brief Title: A Bioequivalence Study of the Fixed Dose Combination Tablets of Canagliflozin and Metformin Extended Release (XR) With Respect to the Individual Components in Healthy Fed Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR103257; 28431754DIA1062 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin; Metformin; Type 2 diabetes mellitus; Bioequivalence; GLUMETZA®
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Experimental): Each participant will receive a single dose of 1 tablet of canagliflozin (CANA), 100 mg, and 4 tablets of metformin extended release (MET XR), 500 mg, administered together under fed conditions.
  Interventions: Drug: Canagliflozin, 100 mg; Drug: Metformin XR, 500 mg
- Treatment B (Experimental): Each participant will receive a single dose of 2 tablets of CANA/MET XR FDC, formulation 1, under fed conditions.
  Interventions: Drug: CANA/MET XR FDC, Formulation 1, 50 mg/1000 mg
- Treatment C (Experimental): Each participant will receive a single dose of 2 tablets of CANA/MET XR FDC, formulation 2, under fed conditions.
  Interventions: Drug: CANA/MET XR FDC, Formulation 2, 50 mg/1000 mg

INTERVENTIONS:
Drug: Canagliflozin, 100 mg — Each tablet contains canagliflozin (CANA) of 100 mg to be taken orally (by mouth).
  Arms: Treatment A
Drug: Metformin XR, 500 mg — Each tablet contains metformin extended release (MET XR), 500 mg, to be taken orally (by mouth).
  Arms: Treatment A
Drug: CANA/MET XR FDC, Formulation 1, 50 mg/1000 mg — Each tablet contains 50 mg of canagliflozin and 1000 mg of metformin HCl granulate, formulation 1, to be taken orally.
  Arms: Treatment B
Drug: CANA/MET XR FDC, Formulation 2, 50 mg/1000 mg — Each tablet contains 50 mg of canagliflozin and 1000 mg of metformin HCl granulate, formulation 2, to be taken orally.
  Arms: Treatment C

SUMMARY:
The purpose of this study is to assess the bioequivalence (similarity of the drug amount in blood among the formulations) of the fixed dose combination (two components combined in one tablet) of canagliflozin and metformin extended release (XR) tablet (dose of 2 X 50 mg/1000 mg) with respect to the individual components of canagliflozin (1 x 100 mg) and metformin XR tablet (4 x 500 mg) in healthy fed participants.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), open-label (physicians and participants know the identity of the assigned treatment), single-center, single-dose, 3-treatment, 3-way crossover (the same medications provided to all participants but in different sequence) study of Fixed Dose Combination (FDC) tablets of canagliflozin (CANA) and metformin extended release (MET XR) in comparison with tablets of individual components. Two Fixed Dose Combinations (FDCs) will be evaluated during the study (two types of tablets). The tablets will be of the same strength (50 mg CANA/1,000 mg MET XR) and will be compared with equal doses of the individual drugs: canagliflozin (1 x 100 mg tablet) and metformin XR (4 x 500 mg tablets). Thus, there will be 3 treatment periods in the study: Treatment A: "Reference" treatment of individual components. Treatment B: CANA/MET XR FDC, formulation 1; and Treatment C: CANA/MET XR FDC, formulation 2. Approximately 42 healthy adult participants will be randomly assigned to 1 of 3 treatments groups, and then each group will receive all three treatments in different sequences (3-way crossover). The study will consist of 3 phases: a Screening Phase of approximately 3 weeks (Days -22 to -2), an Open-Label Treatment Phase consisting of 3 single-dose Treatment Periods of 5 days each (Days -1 through 4) separated by a washout of 10 to 14 days between Day 1 of each Treatment Period, and a Follow-up Phase occurring 7 to 10 days after the last study-related procedure on Day 4 of Treatment Period 3. The total duration of the study will be about 70 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document indicating they understand the purpose of the study and procedures
* Must have a body mass index (BMI) of between 18 and 30 kg/m², inclusive
* Must have a body weight of not less than 50 kg
* Must have a blood pressure between 90 and 140 mmHg inclusive, systolic, and no higher than 90 mmHg diastolic at screening
* Must have normal renal function and no evidence of kidney damage (including abnormalities in blood or urine tests)

Exclusion Criteria:

* History of or current clinically significant medical illness
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements)
* History of clinically significant allergies, especially known hypersensitivity or intolerance to drugs or lactose
* Known allergy to heparin or history of heparin induced thrombocytopenia
* Donated blood or blood products or had substantial loss of blood within 3 months before screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of canagliflozin following the single dose of drug administration | Day 1 to Day 2 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose); Day 3 (48 hour); and Day 4
  Plasma concentrations of canagliflozin are used to evaluate how long canagliflozin stays in the body.
Plasma concentration of metformin following the single dose of drug administration | Day 1 to Day 2 (predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, and 30 hours postdose); and Day 3 (36 hours)
  Plasma concentrations of metformin are used to evaluate how long it stays in the body.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to Day 10 of the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States